CLINICAL TRIAL: NCT07158866
Title: Dance On 50+: Effects of a Dance Program on Physical and Psycho-emotional Health
Brief Title: DanceOn50+: Effects of a Dance Program on Physical and Psycho-emotional Health
Acronym: Dance On 50+
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CEFADE 31_2023
Record Dates: First submitted 2025-02-11; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-07

CONDITIONS: Physical Activity; Physical Fitness; Well Being
Keywords: Active aging; Physical fitness; Cognitive health; Psycho-emotional health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Physical Activity Intervention (Dance Classes and Multicomponent exercises)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ballroom dance Group (Experimental)
  Interventions: Behavioral: Ballroom Dance
- Multicomponent Exercise Group (Experimental)
  Interventions: Behavioral: Multicomponent Exercise
- control group (No Intervention): Participants from the control group will participate in all assesments moments and will be asked to maintain their usual activities. At the end of intervention period, the contol group will be invited to participate in a physical activity program.

INTERVENTIONS:
Behavioral: Ballroom Dance — The intervention will involve twice-weekly dance sessions, lasting 45 minutes each, for 6 months. Each session will include:
  1. Rhythmic warm-up with music.
  2. Combination of aerobic, resistance, and coordination exercises.
  3. Technical development and learning of dance routines.
  4. Cool down with free-body movements to slow music.
  Arms: Ballroom dance Group
Behavioral: Multicomponent Exercise — The Multicomponent Exercise intervention will target several physical fitness components simultaneously, including strength, balance, and aerobic fitness. The program will consist of twice-weekly sessions, each lasting 45 minutes, for 6 months. Each session will include:
  1. Warm-up with light stretching and joint mobility exercises.
  2. Balance exercises
  3. Strength training exercises
  4. Aerobic exercises
  5. Cool down with flexibility and relaxation exercises.
  Arms: Multicomponent Exercise Group

SUMMARY:
Aging is associated with a decline in physical and cognitive function affecting autonomy and the ability to perform daily living activities. Interventions aiming the promotion of healthy aging and life-long learning are required to improve physical and cognitive health in a social context.

Dance is a cultural and physical activity that can be well adapted for older adults. Dance might counteract physical and cognitive functional decline and promotes social and emotional interactions. Importantly, dance can be individually adjusted in terms of physical fitness and cultural background. However, to date, there is a lack of research on the effects of a dance intervention with older adults setting to promote healthy aging and lifelong learning. Thus, this research project aims to explore the impact of a dance-based intervention with older adults from the community on physical, cognitive and psycho-emotional health while simultaneously generating inclusive artistic experiences and lifelong learning opportunities.

The study includes a quantitative quasi-experimental design. The study sample consists of healthy individuals from the community aged ≥ 50 years recruited through community programs and social media platforms. Those who agree to participate will be informed of the project objectives and procedures. Participation in the study is voluntary, and all participants will be required to sign a voluntary informed consent form.

Participants will be assigned to a dance training group, Multicomponent Exercise Group or the control group (no intervention). Outcomes will be measured using the Astrand Cycle Ergometer Submaximal Test, Open Circuit Pirometer Technique, Battery Senior Fitness Test, Isokinetic Dynamometer and Handgrip Dynamometer to assess physical fitness, Accelerometer, and Pittsburgh Sleep Quality Index to assess physical activity, sedentary behaviour, and sleep; psychoemotional questionnaires validated on Portuguese subjects to assess psychoemotional variables; tape measure and bioeletric impedance balance to assess body composition; digital sphygmomanometer and spirometry to assess cardiovascular and respiratory function; neurocognitive and psychological tests to assess cognitive function; and electroencephalography to assess electrophysiology.

DETAILED DESCRIPTION:
The benefits of a dance intervention for Older Adults (OA) may go beyond those associated with PA. A dance program for OA showed improvements in strength, aerobic endurance, flexibility, motor agility/dynamic balance and suggested that PA that endorses cognitive stimulation is more effective in promoting psychological benefits. Dancing for OA based on choreographies, increased volumes in brain regions related to higher cognitive processes including, working memory and attention. Dancing stimulates a large number of physiological processes at the same time: spatial orientation, movement coordination, balance, endurance, interaction and communication, counteracting age-related declines in brain structure. An elegant review suggests the protective effect of a dance intervention on cognition in OA and states that the possibility of adapting intensity and style to suit possible physical limitations makes this activity very suitable for OA. There are also suggestions that, even in older intermediate-level dancer, the practice of social dance might positively influence body composition and also increase fitness performance, memory and anxiety.

Dance requires the synergy of physical and cognitive faculties, using the body to communicate and create an aesthetic form of artistic expression, promoting social and emotional interactions. Dancing improves mental wellbeing and fitness, promoting a sense of community, intimacy, enjoyment and self-fulfillment. Krekula's interviews with OA show that age can be challenged through dance, with the ageing body viewed as a 'source of passion', rather than problematic and people feeling younger, which correlates with higher subjective wellbeing.

Although dance can promote health-related benefits in OA, it is recognized that the few studies in the field seem very heterogonous regarding the trial designs, characteristics of the interventions, outcomes assessments, and methodological quality. Additionally, there are a lack of studies reporting the effects of different styles (i. e. creative, ballroom, traditional dances and others) and its intensity on physical function, particularly in OA. From our knowledge, there are limited studies, on OA, characterizing:

1. the intensity of ballroom dance sessions;
2. physical and cardiorespiratory adaptative responses induced by a ballroom dance program;
3. cognitive and psycho-emotional benefits induced by a ballroom dance program. Therefore, in order to recommend dance as a health promoter intervention for OA, it is urgent to evaluate health-related outcomes of a structured dancing community program.

The present project is a community-based intervention. The majority of existing studies on dance focus on specific populations that have been screened for certain conditions, whereas we will encompass a general population of older adults. To our knowledge, there is a lack of information regarding dance sessions characterization, as well as the health outcomes that a group dance intervention can possibly modulate, including cognitive, physical function and psycho-emotional variables. Therefore, the two main research questions behind this project are:

1. What physical exercise intensity can be achieved during dance sessions for older adults?
2. Can a dance-based intervention positively impact physical, cognitive and psycho-emotional health-related outcomes? To address these questions, the present project aims to characterize dance sessions and explore the impacts of a group dance intervention for older adults within the community, with a focus on simultaneously promoting physical, functional, and cognitive capacities. To provide a comprehensive analysis, comparisons will be made with a control group and a multicomponent exercise group, which is one of the most extensively studied exercise interventions for older adults The research will adopt a quantitative quasi-experimental design and will take place in the metropolitan region of Porto, Portugal. The participant pool will include healthy individuals aged 50 and above, recruited through community programs, local municipalities, health centers, and social media platforms via phone calls and informational brochures. Those who consent to participate will be thoroughly informed about the aims and methods of the study. Participation will be voluntary, and all participants will be asked to sign an informed consent form before taking part in the study.

Participants will be randomly assigned to one of three groups:

1. Dance On group (dance intervention).
2. Multicomponent Exercise group (multicomponent physical training).
3. Control group (no engagement in planned physical activities). Screening will be carried out using a comprehensive questionnaire, collecting socio-demographic and health-related information to ensure that participants meet the inclusion and exclusion criteria for each group.

ELIGIBILITY:
Inclusion criteria:

* 50 years or over;
* informed consent signed;
* not be institutionalized;
* not participating in any type of physical exercise program in the last 3 months.

Exclusion criteria:

* absence of dementia;
* unstable cardiovascular disease or musculoskeletal dysfunction that makes participation in moderate-intensity exercises impossible

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Psychological testing (Depression) - GDS | Baseline, 6 months
  The Geriatric Depression Scale (GDS, short version) will be used to assess depressive symptoms. The Geriatric Depression Scale (GDS), short version, is a self-report instrument developed specifically to screen for depressive symptoms in older adults. The short version consists of 15 yes/no questions, selected from the original 30-item version, and is designed to minimize the influence of somatic symptoms that may overlap with physical ageing processes. Its simplicity and clarity make it especially suitable for older populations, including those with mild cognitive impairments.
  This tool has been widely validated across various settings and cultures, demonstrating good sensitivity and specificity for detecting clinically relevant depressive symptoms in the elderly. Scores range from 0 to 15, with higher scores indicating greater depressive symptomatology. Cut-off points commonly used are: 0-4 (normal), 5-8 (mild depression), 9-11 (moderate depression), and 12-15 (severe depression).
  In
Psychological testing (Anxiety) - EADS-21 | Baseline, 6 months
  Anxiety symptoms will be assessed using the Hamilton Anxiety Rating Scale (HARS), also known as Escala de Ansiedade de Hamilton (EADS) in its Portuguese version. The HARS is a clinician-administered scale that evaluates the severity of anxiety symptoms across psychological and physical domains. It is widely recognized for its high reliability and validity, and is used in both clinical and research settings.
  The scale consists of 14 items that assess various aspects of anxiety, such as tension, fears, insomnia, cognitive impairment, somatic complaints, and autonomic symptoms. Each item is rated on a 5-point Likert scale, ranging from 0 (absent) to 4 (severe).
  The total score can range from 0 to 56, with higher scores indicating more severe levels of anxiety. The commonly used classification is as follows:
  0-17: Mild anxiety 18-24: Moderate anxiety 25-56: Severe anxiety
Peak oxygen uptake (VO2 peak) | Baseline, 6 months
  The Astrand Cycle Ergometer - This sub-maximal test with incremental protocol and performed on a ergometer, standard an open-circuit spirometer technique (Cosmed K5b2, Cosmed, Rome, Italy) will be used.
Lower-body strength and power | Baseline, 6 months
  The knee extensors and flexors will be evaluated using an isokinetic dynamometer at two different angular velocities: 60°/s and 180°/s.
Physical-Functional Fitness (strength of the lower and upper body) | Baseline, 3 months, 6 months
  Physical-functional fitness is going to be measured via the Senior Fitness Test (SFT). This physical battery includes lower and upper-body strength (30-second chair stand and 30-second arm curl tests, respectively), agility/dynamic balance (8-foot up-and-go test), aerobic endurance (six-minute walk test) and lower and upper-body flexibility (chair sit-and-reach and back scratch tests, respectively). The chair stand test to assess the strength of the lower body, counting the number of repetitions made in 30s. And the arm curl test to assess the strength on the upper body, using a 3lb (women) and 5lb (men) dumbbell, counting the number of repetitions made in 30s.
Physical-Functional Fitness (agility/dynamic balance) | Baseline, 3 months, 6 months
  Physical-functional fitness is going to be measured via the Senior Fitness Test (SFT). This physical battery includes lower and upper-body strength (30-second chair stand and 30-second arm curl tests, respectively), agility/dynamic balance (8-foot up-and-go test), aerobic endurance (six-minute walk test) and lower and upper-body flexibility (chair sit-and-reach and back scratch tests, respectively). The stand up, walk 8-foot distance (2,44 meters), turn the cone marker around and return to the seated position. The time, in seconds, necessary to complete this test will be registered.
Physical-Functional Fitness (aerobic endurance) | Baseline, 3 months, 6 months
  Physical-functional fitness is going to be measured via the Senior Fitness Test (SFT). This physical battery includes lower and upper-body strength (30-second chair stand and 30-second arm curl tests, respectively), agility/dynamic balance (8-foot up-and-go test), aerobic endurance (six-minute walk test) and lower and upper-body flexibility (chair sit-and-reach and back scratch tests, respectively). The stand up, walk 8-foot distance (2,44 meters), turn the cone marker around and return to the seated position. The time, in seconds, necessary to complete this test will be registered.
Physical-Functional Fitness (flexibility of the lower and upper-body) | Baseline, 3 months, 6 months
  Physical-functional fitness is going to be measured via the Senior Fitness Test (SFT). This physical battery includes lower and upper-body strength (30-second chair stand and 30-second arm curl tests, respectively), agility/dynamic balance (8-foot up-and-go test), aerobic endurance (six-minute walk test) and lower and upper-body flexibility (chair sit-and-reach and back scratch tests, respectively). The chair sit-&-reach test to assess the flexibility of the lower-body, measured in cm. And The back scratch test to assess flexibility on the upper-body, measured in cm.
Handgrip strength | Baseline, 3 months, 6 months
  The handgrip strength will be measured with a Jamar Plus + Digital hand dynamometer (Sammons Preston Inc., Bolingbrook, Illinois, USA). Measurements will be carried out following the American Society of Hand Therapists recommendations, and each participant will perform three attempts with a pause of 1 min between them. Three attempts will be made for each hand, using the maximum value of the three registers.
Sociodemographic Assessments | Baseline
  Age (years), academic level (primary, secondary, bachelor, master, PhD), civil status (married, separated, widow, single, others), number of medications, diagnosed diseases.
Body mass | Baseline, 6 months
  Body mass (kg) will be analyzed with bioimpedance balance.
World Health Organization Quality of Life - WHOQOL - BREF | Baseline, 6 months
  To assess participants perceived quality of life, the World Health Organization Quality of Life questionnaire (WHOQOL-BREF) will be used. This validated instrument consists of 26 items that measure four key domains: Physical Health, Psychological Health, Social Relationships, and Environment. Each item is rated on a 5-point Likert scale, and scores for each domain are calculated by summing specific items, then transforming the raw scores into a scale from 0 to 100, where higher scores indicate better perceived quality of life.
Life Satisfaction - SWLS | Baseline, 6 months
  To assess overall life satisfaction, the Satisfaction with Life Scale (SWLS) will be administered. This instrument includes 5 items that reflect a global evaluation of an individual's life according to their own criteria and values. In this study, responses will be rated on a 6-point Likert scale ranging from 0 ("Strongly disagree") to 5 ("Strongly agree"), resulting in a total score ranging from 0 to 25. Higher scores indicate greater satisfaction with life. Interpretation of total scores typically follows these cut-offs: 0-4 (Extremely dissatisfied), 5-9 (Dissatisfied), 10-14 (Slightly dissatisfied), 15 (Neutral), 16-19 (Slightly satisfied), 20-22 (Satisfied), and 23-25 (Extremely satisfied).
Loneliness - UCLA-16 | Baseline, 6 months
  To assess perceived social isolation, this study will use the Portuguese-adapted version of the UCLA Loneliness Scale comprising 16 items. This version was culturally and linguistically validated for the Portuguese population, particularly in older adults, ensuring conceptual equivalence while excluding or modifying items less relevant in this context. Each item is rated on a 4-point Likert scale ranging from 1 ("Never") to 4 ("Often"). Total scores range from 16 to 64, with higher scores indicating greater perceived loneliness. The scale assesses key dimensions of loneliness, including feelings of social disconnectedness, lack of companionship, and emotional isolation.
Positive and Negative Affect - PANAS | Baseline, 6 months
  To evaluate affective states, the study will use the Positive and Negative Affect Schedule (PANAS), a validated self-report instrument measuring two distinct dimensions of mood: Positive Affect (PA) and Negative Affect (NA). The PANAS consists of 20 items, with 10 items assessing PA-enthusiastic, interested, alert, inspired, determined, attentive, active, proud, excited, and strong-and 10 items assessing NA-distressed, upset, guilty, scared, hostile, irritable, ashamed, nervous, jittery, and afraid. Participants rate how much they have experienced each emotion over a specified time frame on a 5-point Likert scale ranging from 1 ("Very slightly or not at all") to 5 ("Extremely"). Scores for each subscale are summed separately, with possible ranges of 10 to 50. Higher PA scores indicate greater positive emotional engagement, while higher NA scores reflect higher levels of distress and negative emotional experience.
Physical Activity | Baseline, 6 months
  Physical Activity will be tested by Accelerometer-based activity monitors GT3X+ Link (ActiGraph)
Sleep Quality - PSQI-PT | Baseline, 6 months
  To assess sleep quality, the study will use the Pittsburgh Sleep Quality Index - Portuguese version (PSQI-PT), a widely validated self-report questionnaire designed to measure sleep quality and disturbances over a one-month period. The PSQI-PT consists of 19 items, which generate seven component scores assessing different dimensions of sleep: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component is scored from 0 to 3, and the sum of these yields a global score ranging from 0 to 21. Higher scores indicate poorer sleep quality, with a commonly used cut-off of >5 to distinguish poor sleepers from good sleepers.
fat-free mass | baseline, months
  fat-free mass (kg), will be analyzed with bioimpedence balance.
fat mass | baseline, 6 months
  fat mass (%) will be analyzed with bioimpedance balance.
BMI - Body Mass Index | baseline, 6 months
  BMI (Kg/m^2) will be analyzed with bioimpedance balance.

SECONDARY OUTCOMES:
Cognitive performance (Memory) | Baseline, 6 months
  Consortium to establish a registry for the Alzheimer's Disease List Test (CERAD), will be used: word list memory; word list recall; and word list recognition. The parameters: total hits and delayed recall hits.
Cognitive performance (Selective recall test) | Baseline, 6 months
  Selective recall test [SRT-List A; parameters: consistent long-term recall, long-term storage, delayed recall, and intrusions] to assess verbal learning and multiple-trial memory.
Cognitive performance (Verbal short-term memory) | Baseline, 6 months
  The Forward Digit Span (DS) test will be used to assess verbal short-term memory. This test is a subtest of the Wechsler Adult Intelligence Scale (WAIS-III).
  The Forward DS test requires participants to repeat a sequence of digits in the same order they were presented, assessing their ability to hold and recall information over a short period.
  The DS score is determined by the maximum number of digits the participant is able to accurately repeat in the correct order. A performance of 5 to 7 digits falls within the normative range. Scores below this range may indicate potential deficits in attention or short-term memory capacity, while scores above may reflect superior cognitive functioning.
Cognitive performance (Inhibition/cognitive flexibility) | Baseline, 6 months
  The Stroop Color and Word Test (parameters: words, colors, and words/colors) will be selected to assess response inhibition/cognitive flexibility.
Cognitive performance (Processing speed) | Baseline, 6 months
  Digit Symbol Substitution Test (DSST, subtest of the Wechsler test of adult intelligence WAIS III) will be used as a measure of high-level information processing speed.
Brain Activity | Baseline, 6 months
  This will be analyzed using an electromyography (EEG) system. All EEG signals will be acquired with the ActiCHamp®, Brain Products,GmbH. With an international 10-20 system with standard 32-channel electrode layout with reference and ground electrodes. The ground will be located on the forehead and the reference will be the Cz channel of the ActiCHamp® equipment. For each participant, the same equipment will be used in all sessions.
Risk of Falls - FRAX | Baseline, 6 months
  Risk of falls will be evaluated through The Fracture Assessment Risk Tool (FRAX).
Perceptions of the experience of participants | 6 months
  Qualitative analysis will be testd with Semi-structured interviews.
Cognitive Performance (Verbal Working Memory) | Baseline, 6 months
  Working memory will be assessed using the Backward Digit Span subtest from the Wechsler Adult Intelligence Scale - Third Edition (WAIS-III). In this task, participants are required to repeat a sequence of digits in the reverse order of their presentation, evaluating their ability to mentally manipulate and retain verbal information. The Backward DS score is defined as the highest number of digits the participant can accurately reproduce in the correct reverse sequence. Performance typically ranges from 3 to 5 digits, based on normative data. Scores below this range may indicate difficulties in working memory or executive functioning, whereas scores above may suggest enhanced cognitive flexibility and working memory capacity.
  Time Frame: Baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: José Magalhães, PhD, Study Director — Faculty of Sport, University of Porto
Locations (1):
- CIAFEL, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No
Data will be produced and stored in accordance with the data protection laws and the University of Porto internal regulations. Data collected by questionnaire and direct observation will be anonymized before storage. The sub-investigator will be the only person with access to the grid that contains the data coding. Data will be stored in the official University of Porto cloud and with a copy on a hard disk that will be in the sub-investigator possession.

REFERENCES:
- [Background] Rodrigues-Krause J, Krause M, Reischak-Oliveira A. Dancing for Healthy Aging: Functional and Metabolic Perspectives. Altern Ther Health Med. 2019 Jan;25(1):44-63. PMID 29428927
- [Background] Vaccaro MG, Izzo G, Ilacqua A, Migliaccio S, Baldari C, Guidetti L, Lenzi A, Quattrone A, Aversa A, Emerenziani GP. Characterization of the Effects of a Six-Month Dancing as Approach for Successful Aging. Int J Endocrinol. 2019 Jun 17;2019:2048391. doi: 10.1155/2019/2048391. eCollection 2019. PMID 31316562
- [Background] 19- Physical Activity Guidelines Advisory Committee, 2018. Physical Activity Guidelines Advisory Committee Scientific Report. Washington, DC: U.S. Department of Health and Human Services
- [Background] Rehfeld K, Luders A, Hokelmann A, Lessmann V, Kaufmann J, Brigadski T, Muller P, Muller NG. Dance training is superior to repetitive physical exercise in inducing brain plasticity in the elderly. PLoS One. 2018 Jul 11;13(7):e0196636. doi: 10.1371/journal.pone.0196636. eCollection 2018. PMID 29995884
- [Background] Wilde NJ, Strauss E, Chelune GJ, Hermann BP, Hunter M, Loring DW, Martin RC, Sherman EM. Confirmatory factor analysis of the WMS-III in patients with temporal lobe epilepsy. Psychol Assess. 2003 Mar;15(1):56-63. doi: 10.1037/1040-3590.15.1.56. PMID 12674724
- [Background] Buschke H, Sliwinski M, Kuslansky G, Lipton RB. Aging, encoding specificity, and memory change in the Double Memory Test. J Int Neuropsychol Soc. 1995 Sep;1(5):483-93. doi: 10.1017/s1355617700000576. PMID 9375233
- [Background] Morris JC, Heyman A, Mohs RC, Hughes JP, van Belle G, Fillenbaum G, Mellits ED, Clark C. The Consortium to Establish a Registry for Alzheimer's Disease (CERAD). Part I. Clinical and neuropsychological assessment of Alzheimer's disease. Neurology. 1989 Sep;39(9):1159-65. doi: 10.1212/wnl.39.9.1159. PMID 2771064
- [Background] Del Rio Joao KA, Becker NB, de Neves Jesus S, Isabel Santos Martins R. Validation of the Portuguese version of the Pittsburgh Sleep Quality Index (PSQI-PT). Psychiatry Res. 2017 Jan;247:225-229. doi: 10.1016/j.psychres.2016.11.042. Epub 2016 Nov 28. PMID 27923147
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] 10- Pocinho, M., Farate, C. & Dias, C., (2010). Validação Psicométrica da Escala UCLA-Lonliness para Idosos Portugueses. Interções. 65-77.
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] 8- World Health Organization. (2021). Obesity and Overweight. Retrieved July 2023 from https://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight
- [Background] 6-Nagata, C. d. A., Hamu, T. C. D. d. S., Neri, S. G. R., Lima, R. M., & Garcia, P. A. (2023). Association between isokinetic strength measures and functional performance in community-dwelling older adults. Fisioterapia e Pesquisa, 30, e22014323en
- [Background] 5- Krekula, C., Pleasure and time in senior dance: bringing temporality into focus in the field of ageing. Ageing and Society, 2020: p. 1-16.
- [Background] Cruz-Ferreira A, Marmeleira J, Formigo A, Gomes D, Fernandes J. Creative Dance Improves Physical Fitness and Life Satisfaction in Older Women. Res Aging. 2015 Nov;37(8):837-55. doi: 10.1177/0164027514568103. Epub 2015 Jan 29. PMID 25651595
- [Background] Krekula C, Arvidson M, Heikkinen S, Henriksson A, Olsson E. On gray dancing: Constructions of age-normality through choreography and temporal codes. J Aging Stud. 2017 Aug;42:38-45. doi: 10.1016/j.jaging.2017.07.001. Epub 2017 Aug 8. PMID 28918820
- [Background] 1- Pais-Ribeiro, J. L., Honrado, A., & Leal, I. (2004). Contribuição Para O Estudo Da Adaptação Portuguesa Das Escalas De Ansiedade , Depressão E Stress ( Eads ) De 21 Itens De Lovibond E Lovibond. Psicologia, Saúde & Doenças, 5(2), 229-239.